CLINICAL TRIAL: NCT05889689
Title: Relationship Smarts Plus and Mind Matters: A Randomized Control Trial of a High School Intervention to Reduce Sexual Risk Behaviors.
Brief Title: Evaluation of an Adolescent Pregnancy Prevention Program; Relationship Smarts+ With Lessons From Mind Matters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Church Inc. (Other)
Collaborators: AMTC & Associates (Unknown); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90AP2700-01-00
Record Dates: First submitted 2023-05-12; First posted 2023-06-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-05

CONDITIONS: Teen Pregnancy; Contraception Behavior; Sexually Transmitted Diseases; Reproductive Health; Sexual Risk Behavior
MeSH Terms: conditions — Contraception Behavior; Sexually Transmitted Diseases | interventions — Single Person

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relationship Smarts Plus & Mind Matters (Experimental): Relationship Smarts Plus (RSP+) is an adolescent pregnancy prevention curriculum that will be combined with lessons from a trauma-coping skills curriculum, Mind Matters (MM).
  Interventions: Behavioral: Relationship Smarts Plus & Mind Matters
- Relationship Smarts Plus (Experimental): Relationship Smarts Plus (RSP+) is an adolescent pregnancy prevention curriculum.
  Interventions: Behavioral: Relationship Smarts Plus alone
- Control Group (Active Comparator): Financial literacy curriculum, Preparing Adolescents for Young Adulthood (PAYA)
  Interventions: Behavioral: Preparing Adolescents for Young Adulthood (PAYA).

INTERVENTIONS:
Behavioral: Relationship Smarts Plus & Mind Matters — 18.5 hours long intervention that combines the Relationship Smarts Plus teen pregnancy prevention curriculum with lessons from the Mind Matters trauma-coping skills curriculum
  Arms: Relationship Smarts Plus & Mind Matters
Behavioral: Relationship Smarts Plus alone — 14-hour-long curriculum that addresses pregnancy prevention within the context of teaching relationship skills for young teens.
  Arms: Relationship Smarts Plus
Behavioral: Preparing Adolescents for Young Adulthood (PAYA). — A financial literacy curriculum
  Arms: Control Group

SUMMARY:
The goal of this randomized control trial (RCT) is to assess an innovative adolescent pregnancy prevention program among youth that are at the highest risk of adolescent pregnancy, to prevent pregnancy and Sexually Transmitted Infections (STIs), including HIV/AIDS in the greater Miami area in Florida. The primary research question it aims to answer is:

(RQ1a): What is the effect of adding 4.5 hours of Mind Matters trauma-coping skills curriculum to the Relationship Smarts Plus curriculum, on rates of unprotected sex among 9th and 10th graders compared to the students receiving only the 14-hour-long Relationship Smarts Plus curriculum? (RQ1b): What is the effect of the 14-hour-long Relationship Smarts Plus curriculum on rates of unprotected sex among 9th and 10th graders compared to the control group receiving only financial literacy? Participants will complete program lessons and complete surveys for data collection.

The RCT will assess behavioral health outcomes and other psychological outcomes at four-time points (baseline, post-program, 3 months, and 12 months)

DETAILED DESCRIPTION:
The intervention combines the pregnancy prevention curriculum, Relationship Smarts Plus (RSP+) with lessons from the trauma coping skills curriculum, Mind Matters (MM). The mental health component was added to assess the importance of mental health as a risk factor for teen pregnancy. Researchers will estimate the effect of Mind Matters (MM) by comparing the RSP+ & MM treatment arm with the RSP+ treatment arm. This answers RQ1a: If MM has an impact, then researchers will answer RQ1b by comparing the RSP+ treatment arm with the control arm. If there's no impact, then RQ1b will be answered by comparing the pooled RSP+ and RSP+ & MM treatment arms with the control arm.

This study is funded through the Personal Responsibility Education Program Innovative Strategies (PREIS), which is administered by the Family and Youth Services Bureau, part of Health and Human Services,

Trinity Church, Miami Gardens, is responsible for site and participant recruitment as well as the implementation of the intervention. Participants are randomized at the classroom level. All control group participants will only receive a financial literacy program.

AMTC & Associates is the external evaluator, The Dibble Institute is the curricula developer.

ELIGIBILITY:
Inclusion Criteria:

For schools to be included in the study:

They have to be located within the greater Miami area.

For individuals:

1. Students enrolled in either 9th,10th, 11th and 12th grade
2. Students who do not have severe cognitive, mental health, or behavioral impairment.
3. Students with Individualized Education Plans who are part of the mainstream classrooms.

Exclusion Criteria:

1. Students who do not consent to be in the study
2. Students who are part of the pilot study
3. Students who have been randomized in a previous cohort of the study
4. Students with an Individualized Education Plan (IEP) who are in restricted placement will not be able to participate in the program as they will not be part of the mainstream classrooms where the program is implemented.
5. Students who have received such a program within the last year will be eligible to participate in the program but will be excluded from statistical analysis to ensure the results are not biased from participation in a similar curriculum.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2250 (Estimated)
Dates: Start 2023-09-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Unprotected sex as measured by 4 items from the survey. The 4 items will be combined to create a binary variable as an indicator of either protected sex or unprotected sex. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of unprotected sex

SECONDARY OUTCOMES:
Unprotected sex as measured by 4 items from the survey. The 4 items will be combined to create a binary variable as an indicator of either protected sex or unprotected sex. | At 3 months after baseline data collection.
  The proportion of youth who, in comparison to the control group, report lower rates of unprotected sex.
Sexual intercourse as measured by a binary indicator asking participants if they ever engaged in sexual intercourse | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of sexual intercourse
Sexual intercourse as measured by a binary indicator asking participants if they ever engaged in sexual intercourse | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of sexual intercourse
Oral sex as measured by a single binary indicator asking participants if they ever engaged in oral sex | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of oral sex
Oral sex as measured by a single binary indicator asking participants if they ever engaged in oral sex | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of oral sex
Sexual Initiation as measured by a 7- item 5 response ordinal scale categorical indicator of when individuals intent to start engaging in different sexual activities | At 3 months and at 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of sexual initiation
Sexual Initiation as measured by a 7- item 5 response ordinal scale categorical indicator of when individuals intent to start engaging in different sexual activities | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report lower rates of sexual initiation
Skills to negotiate abstinence & resist pressure to have sex measured by a 10-item scale on a 5-point scale showing how confident they are in answering each of the 10 items. A score will be calculated by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report they have the skills to negotiate abstinence and resist pressure to have sex.
Skills to negotiate abstinence & resist pressure to have sex measured by a 10-item scale on a 5-point scale showing how confident they are in answering each of the 10 items. A score will be calculated by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report they have the skills to negotiate abstinence and resist pressure to have sex.
Intent to use condoms as measured by a binary indicator that asks participants if they will use condoms and other contraceptives | At 3 months and at 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report intent to consistently use condoms.
Intent to use condoms as measured by a binary indicator that asks participants if they will use condoms and other contraceptives | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report intent to consistently use condoms.
Knowledge of HIV/STIs as measured by 8-item True/False/Unsure responses to survey items. Items will be scored as 1 if correct & 0 if incorrect. Composite scores of correct items will be calculated. Scores range from 0 to 8 | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher knowledge of HIV/STIs.
Knowledge of HIV/STIs as measured by 8-item True/False/Unsure responses to survey items. Items will be scored as 1 if correct & 0 if incorrect. Composite scores of correct items will be calculated. Scores range from 0 to 8 | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher knowledge of HIV/STIs.
Future-oriented goals as measured by a 10-item 6-point response scale, respondents will show how much they agree or disagree with each of the 10 statements. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report having future-oriented goals
Future-oriented goals as measured by a 10-item 6-point response scale, respondents will show how much they agree or disagree with each of the 10 statements. A score will be calculated for each of the respondents by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report having future-oriented goals
Healthy life skills measured by a 12-item 6-point response scale, respondents will show how much they agree or disagree with each of the 12 items. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more health life skills
Healthy life skills measured by a 12-item 6-point response scale, respondents will show how much they agree or disagree with each of the 12 items. A score will be calculated for each of the respondents by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more health life skills
Awareness of healthy relationships as measured by a 10-item 6-point response scale, respondents will show how much they agree or disagree with each of the 10 statements. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher awareness of healthy relationships
Awareness of healthy relationships as measured by a 10-item 6-point response scale, respondents will show how much they agree or disagree with each of the 10 statements. A score will be calculated for each of the respondents by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher awareness of healthy relationships
General communication skills as measured by a 7-item scale on a 5-point scale, respondents will show how much they agree or disagree with each of the 7 statements. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more communication skills
General communication skills as measured by a 7-item scale on a 5-point scale, respondents will show how much they agree or disagree with each of the 7 statements. A score will be calculated for each of the respondents by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more communication skills
Parent/guardian communication about sex measured by a 6-item scale on a 5-point scale, respondents will show how confident they are in answering each of the 6 items. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more communication skills
Parent/guardian communication about sex measured by a 6-item scale on a 5-point scale, respondents will show how confident they are in answering each of the 6 items. A score will be calculated for each of the respondents by averaging their responses. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more communication skills
Conflict resolution skills as measured using 8 items on a 5-point scale, respondents will show how confident they are in answering each of the 8 statements. A score will be calculated for each of the respondents by averaging their responses. | At 3 months and at 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more conflict resolution skills
Conflict resolution skills as measured using 8 items on a five-point response scale, respondents will show how confident they are in answering each of the 8 statements. A score will be calculated for each of the respondents by averaging their responses. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report more conflict resolution skills
Resilience as measured by the Connor-Davidson Resilience Scale (CD-RISC). A 5 point rating of how participants have felt over the past month. Scores range from 0-4. An average score will be calculated. | At 12 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher resiliency
Resilience as measured by the Connor-Davidson Resilience Scale (CD-RISC). A 5 point rating of how participants have felt over the past month. Scores range from 0-4. An average score will be calculated. | At 3 months after baseline data collection
  The proportion of youth who, in comparison to the control group, report higher resiliency

CONTACTS AND LOCATIONS:
Locations (1):
- Trinity Church Inc, Miami Gardens, Florida, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share Individual Participant Data with other researchers